CLINICAL TRIAL: NCT03137147
Title: Intervention for Sleep and Pain in Youth: A Feasibility Study of Cognitive-Behavioral Intervention
Brief Title: Intervention for Sleep and Pain in Youth
Acronym: I-SPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Emily Law, Assistant Professor, Anesthesiology & Pain Medicine, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000002
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Headache Disorders; Migraine Disorders; Insomnia
Keywords: pediatric; children; adolescent; sleep; pain; cognitive-behavioral therapy
MeSH Terms: conditions — Headache Disorders; Migraine Disorders; Sleep Initiation and Maintenance Disorders; Pain | interventions — Methods; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive-Behavioral Therapy (Other): Intervention for Sleep and Pain in Youth, a 7-session cognitive-behavioral therapy intervention for co-morbid insomnia and headache
  Interventions: Behavioral: Intervention for Sleep and Pain in Youth

INTERVENTIONS:
Behavioral: Intervention for Sleep and Pain in Youth — See arm description.
  Other Names: Hybrid cognitive behavioral therapy for insomnia and headache

SUMMARY:
This study tests the feasibility, acceptability, and preliminary efficacy of a seven-session cognitive-behavioral therapy intervention to treat sleep and pain problems in youth ages 11-17 with co-morbid headache and insomnia.

DETAILED DESCRIPTION:
Cognitive-behavioral interventions have been developed to treat childhood insomnia and childhood headache. In this study, we have combined strategies from these interventions into a single, seven-session protocol to treat sleep and pain problems in youth with co-morbid headache and insomnia. In this single-arm pilot study, we will test the feasibility, acceptability, and preliminary efficacy of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* youth age 11-17 years
* chronic headache and insomnia symptoms for the past 3 months as determined on screening interview with youth and parent.

Exclusion Criteria:

* youth and parent do not read or speak English
* youth with active suicidal ideation or psychosis
* youth with diagnosis of a comorbid serious health condition (e.g., cancer, diabetes)
* youth with severe cognitive impairment
* youth with another primary sleep disorder (e.g., sleep apnea, narcolepsy) or an unusual sleep/wake schedule or circadian rhythm disorder.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Delivery: Number of Completed Intervention Visits | 6-12 weeks
  Number of completed intervention visits
Feasibility of Intervention Delivery: Recruitment/Enrollment Rate | 6-12 weeks
  Recruitment/Enrollment Rate

SECONDARY OUTCOMES:
Treatment Acceptability and Satisfaction: Treatment Evaluation Inventory Short Form | 3 months
  9-item self-report measure of treatment acceptability and satisfaction, scores range from 9-45, higher scores indicate greater treatment acceptability
Insomnia Severity Index | 3 months
  7-item self-report measure of insomnia severity and impact, scores range from 0-28 with higher scores indicating greater insomnia symptoms.
Adolescent Sleep Wake Scale | Past 4 weeks
  28-item measure of subjective sleep quality, scores range from 28-168, higher scores indicate poorer sleep quality
Pain Questionnaire | Past 2 weeks
  Assesses pain frequency, intensity, onset, and duration.
Child Activity Limitations Interview | Past month
  Assesses pain-related disability

CONTACTS AND LOCATIONS:
Overall Officials: Emily Law, PhD, Principal Investigator — University of Washington & Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palermo TM, Beals-Erickson S, Bromberg M, Law E, Chen M. A Single Arm Pilot Trial of Brief Cognitive Behavioral Therapy for Insomnia in Adolescents with Physical and Psychiatric Comorbidities. J Clin Sleep Med. 2017 Mar 15;13(3):401-410. doi: 10.5664/jcsm.6490. PMID 27923435
- [Background] Eccleston C, Palermo TM, Williams AC, Lewandowski Holley A, Morley S, Fisher E, Law E. Psychological therapies for the management of chronic and recurrent pain in children and adolescents. Cochrane Database Syst Rev. 2014 May 5;2014(5):CD003968. doi: 10.1002/14651858.CD003968.pub4. PMID 24796681
- [Background] Fales J, Palermo TM, Law EF, Wilson AC. Sleep outcomes in youth with chronic pain participating in a randomized controlled trial of online cognitive-behavioral therapy for pain management. Behav Sleep Med. 2015;13(2):107-23. doi: 10.1080/15402002.2013.845779. Epub 2014 Jan 31. PMID 24484373
- [Background] Palermo TM, Law E, Churchill SS, Walker A. Longitudinal course and impact of insomnia symptoms in adolescents with and without chronic pain. J Pain. 2012 Nov;13(11):1099-106. doi: 10.1016/j.jpain.2012.08.003. Epub 2012 Sep 30. PMID 23031311
- [Background] Palermo TM, Wilson AC, Lewandowski AS, Toliver-Sokol M, Murray CB. Behavioral and psychosocial factors associated with insomnia in adolescents with chronic pain. Pain. 2011 Jan;152(1):89-94. doi: 10.1016/j.pain.2010.09.035. Epub 2010 Oct 27. PMID 21030151
- [Derived] Law EF, Wan Tham S, Aaron RV, Dudeney J, Palermo TM. Hybrid Cognitive-Behavioral Therapy Intervention for Adolescents With Co-Occurring Migraine and Insomnia: A Single-Arm Pilot Trial. Headache. 2018 Jul;58(7):1060-1073. doi: 10.1111/head.13355. PMID 30152164